CLINICAL TRIAL: NCT04116580
Title: Efficacy of Oral Tolerance Induction to Raw Apple Using an Ultra Rush Protocol in 28 Rosacea Allergic Patients
Brief Title: Efficacy of Oral Tolerance Induction to Raw Apple
Acronym: RAAP
Status: Completed | Type: Observational
Sponsor: Michel Bouvier (Network)
Collaborators: Polyclinique du Beaujolais (Unknown); Clinique Charcot (Unknown)
Responsible Party: Sponsor-Investigator, Michel Bouvier, Principal Investigator, Centre d'Allergologie du Beaujolais
Organization: Centre d'Allergologie du Beaujolais (Network)
Other Study IDs: Apple CAB 1 - 2019
Record Dates: First submitted 2019-08-11; First posted 2019-10-04 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-10

CONDITIONS: Oral Allergic Syndrome; Allergic Reaction Caused by Food (Disorder)
Keywords: Food Allergy; Apple Allergy; Oral Allergic Syndrome; Ultra-Rush; Tolerance induction; Cross-Allergy
MeSH Terms: conditions — Food Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Allergic patients to raw apple and birch: Single-group studies about 28 patients allergic to birch and no longer eating raw rosaceae for at least 6 months. Patients brought back into contact with this family of fruits via the raw golden apple according to an Ultra-Rush protocol.
  Interventions: Other: RAAP - for Raw Apple in connection with re-contact with the raw apple according to an Ultra-Rush protocol

INTERVENTIONS:
Other: RAAP - for Raw Apple in connection with re-contact with the raw apple according to an Ultra-Rush protocol

SUMMARY:
The aim of the study was to describe an intensive ultra rush (UR) protocol of raw Golden apple (RGA) reintroduction in 28 in-patients, show the protocol's tolerance and the patients' follow-up at 2 months and 1 year. Patients with oral allergic syndrome (OAS) having resulted in raw fruits eviction were admitted to day hospital between June 1 2016 and October 31 2017.

DETAILED DESCRIPTION:
The aim of this study was to describe an intensive ultra rush (UR) protocol of raw Golden apple (RGA) reintroduction in 28 in-patients, show the protocol's tolerance and the patients' follow-up at 2 months and 1 year. Patients with oral allergic syndrome (OAS) having resulted in raw fruits eviction were admitted to day hospital between June 1 2016 and October 31 2017.

Methods : Patients were included during the first consultation, UR was performed with RGA in day hospital performed in two institutions, the Charcot clinic and the polyclinic of Beaujolais.

Starting with 1 gram (g) of food, then by regularly doubling dose from 2g to 128g, to reach a 255g cumulative dose in a 3 hour period.

During the the post hospitalization period, patients back home had to eat ½ RGA a day during one month, then 1 RGA a day during one month, together with other rosacea fruits resumption at the end of the 5th week if UR were performed between April 15th and July 15th. A synthesis consultation was made at two months and a telephone interview at one year.

ELIGIBILITY:
Inclusion Criteria:

* No longer eat raw rosacea for at least 6 months due to oral allergic syndrome
* With allergic rhinitis or asthma due to betulaceae pollen (SPT+ and/or IgE + to Bet v 1 > 0,10 kUA/L)
* With reduced quality of life

Exclusion Criteria:

* With severe allergic reaction to rosacea (>Grade 3 according to Ring and Messmer's classification)
* Pregnant woman
* Uncontrolled asthma (FEV1 < 70%)
* Immunosuppressed patient or having malignant disease, current infectious disease, or serious cardiovascular disease
* Opposed to use data

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Food-Pollen Allergic patients aged 10 years and more, allergic to birch pollen and not eating any more rosacee for at least 6 months
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
Patients' tolerance to Golden apple re-consumption according to a Visual Analogue Scale (VAS) | [Time Frame: Day 1]
  Evaluation of the patients' tolerance to apple re-consumption was made during the ultra-rush protocol according to a scale inspired by the Hansen et al. classification, but the VAS used was graduated from 0 to 10 (and not from 0 to 3). This scale was enhanced with a three-color rule: the scale measured 3 levels of Oral Allergic Syndrome (OAS) severity: with no or mild side effects associated with the green color (0 to 3 on the scale), with moderate side effect associated with the orange color (4 to 6 on the scale) defined as moderate OAS (limited to oral cavity), and with severe side effect associated with red color (7 to 10 on the scale) defined as severe OAS (oral cavity together with systemic symptoms).
  Green color corresponds to good tolerability, orange color to mixed results, and red color is correlated to poor tolerability.

SECONDARY OUTCOMES:
Ultra-Rush incidence on blood pressure constants (in mmHg) | [Time Frame: Day 1]
  Measurement of blood pressure constants during Ultra-Rush
Ultra-Rush incidence on pulse rate (in bpm) | [Time Frame: Day 1]
  Measurement of pulse in beats per minute during Ultra-Rush
Ultra-Rush incidence on peak-flow (in liters/mn) | [Time Frame: Day 1]
  Measurement of peak-flow in liters per minute during Ultra-Rush
Procedure's safety on side effects according to a Visual Analogue Scale (VAS) | [Time Frame: Day 1]
  Measurement of side effects during Ultra-Rush (UR) and for the next two months according to the Visual Analogue Scale (VAS) used for the study.
  The 0-10 graduated scale was enhanced with a three-color rule: the scale measured 3 levels of Oral Allergic Syndrome (OAS) severity: with no or mild side effects (green color), with moderate side effect (orange color), and with severe side effect (red color).
  During UR, side effects intensity was evaluated on the VAS at each UR step. After UR and for the next two months, patients recorded daily the side effects on a notebook, using the same tool. These records were transcribed in the patients medical file by investigator.
Tolerance of apple re-consumption on a daily basis during the 2 months following ultra-rush | [Time Frame: Day 1]
  Evaluation of the tolerance by means of visual scale with 3 levels of stringency: without side effects (associated with the green color), with moderate side effect (associated with the orange color) and with severe side effect (associated with red color)
Tolerance of apple and other raw rosacea re-consumption two months post- Ultra-Rush for patients treated between mid-April and mid-July, according to a Visual Analogue Scale (VAS) | [Time Frame: Day 1]
  Tolerance was evaluated at the two months post Ultra-Rush visit, using the VAS. The 0-10 graduated scale was enhanced with a three-color rule: the scale measured 3 levels of Oral Allergic Syndrome (OAS) severity: with no or mild side effects (green color), with moderate side effect (orange color), and with severe side effect (red color).
Number of participants eating rosacea with no or mild OAS at 1 year | [Time Frame: Day 1]
  During a specific interrogation in a telephone interview
Biological sensitization profile of patients included | [Time Frame: Day 1]
  With an initial biological assessment to measure specific: Immunoglobulin E (IgE) apple; rBet v 1 (PR 10 protein); rBet v 2 (profilin protein) et rPru p 3 (lipid transfer protein)

CONTACTS AND LOCATIONS:
Overall Officials: Bouvier Michel, MD, Principal Investigator — Centre d' Allergologie du Beaujolais

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nucera E, Aruanno A, Lombardo C, Patriarca G, Schiavino D. Apple desensitization in two patients with PR-10 proteins allergy. Allergy. 2010 Aug;65(8):1060-1. doi: 10.1111/j.1398-9995.2009.02275.x. Epub 2009 Dec 3. No abstract available. PMID 19958318
- [Background] Kopac P, Rudin M, Gentinetta T, Gerber R, Pichler Ch, Hausmann O, Schnyder B, Pichler WJ. Continuous apple consumption induces oral tolerance in birch-pollen-associated apple allergy. Allergy. 2012 Feb;67(2):280-5. doi: 10.1111/j.1398-9995.2011.02744.x. Epub 2011 Nov 10. PMID 22070352
- [Background] Werfel T, Asero R, Ballmer-Weber BK, Beyer K, Enrique E, Knulst AC, Mari A, Muraro A, Ollert M, Poulsen LK, Vieths S, Worm M, Hoffmann-Sommergruber K. Position paper of the EAACI: food allergy due to immunological cross-reactions with common inhalant allergens. Allergy. 2015 Sep;70(9):1079-90. doi: 10.1111/all.12666. Epub 2015 Jul 7. PMID 26095197
- [Background] Bouvier M; Van der Brempt X; Nosbaum A; Cordier JM; Nicolas JF; Berard F. Induction of oral tolerance in allergy to rosaceae. Revue Française d'Allergologie (54): 127-133, 2014
- [Background] Muraro A, Werfel T, Hoffmann-Sommergruber K, Roberts G, Beyer K, Bindslev-Jensen C, Cardona V, Dubois A, duToit G, Eigenmann P, Fernandez Rivas M, Halken S, Hickstein L, Host A, Knol E, Lack G, Marchisotto MJ, Niggemann B, Nwaru BI, Papadopoulos NG, Poulsen LK, Santos AF, Skypala I, Schoepfer A, Van Ree R, Venter C, Worm M, Vlieg-Boerstra B, Panesar S, de Silva D, Soares-Weiser K, Sheikh A, Ballmer-Weber BK, Nilsson C, de Jong NW, Akdis CA; EAACI Food Allergy and Anaphylaxis Guidelines Group. EAACI food allergy and anaphylaxis guidelines: diagnosis and management of food allergy. Allergy. 2014 Aug;69(8):1008-25. doi: 10.1111/all.12429. Epub 2014 Jun 9. PMID 24909706
- [Background] Mauro M, Russello M, Incorvaia C, Gazzola G, Frati F, Moingeon P, Passalacqua G. Birch-apple syndrome treated with birch pollen immunotherapy. Int Arch Allergy Immunol. 2011;156(4):416-22. doi: 10.1159/000323909. Epub 2011 Aug 10. PMID 21832831
- [Background] Incorvaia C, Ridolo E, Mauro M, Russello M, Pastorello E. Allergen immunotherapy for birch-apple syndrome: what do we know? Immunotherapy. 2017 Nov;9(15):1271-1278. doi: 10.2217/imt-2017-0040. PMID 29130794
- [Background] Hansen KS, Khinchi MS, Skov PS, Bindslev-Jensen C, Poulsen LK, Malling HJ. Food allergy to apple and specific immunotherapy with birch pollen. Mol Nutr Food Res. 2004 Nov;48(6):441-8. doi: 10.1002/mnfr.200400037. PMID 15508179
- [Background] Kinaciyan T, Jahn-Schmid B, Radakovics A, Zwolfer B, Schreiber C, Francis JN, Ebner C, Bohle B. Successful sublingual immunotherapy with birch pollen has limited effects on concomitant food allergy to apple and the immune response to the Bet v 1 homolog Mal d 1. J Allergy Clin Immunol. 2007 Apr;119(4):937-43. doi: 10.1016/j.jaci.2006.11.010. Epub 2007 Jan 3. PMID 17204315
- [Background] Scala E, Abeni D, Guerra EC, Locanto M, Pirrotta L, Meneguzzi G, Giani M, Asero R. Cosensitization to profilin is associated with less severe reactions to foods in nsLTPs and storage proteins reactors and with less severe respiratory allergy. Allergy. 2018 Sep;73(9):1921-1923. doi: 10.1111/all.13501. Epub 2018 Jun 22. No abstract available. PMID 29885248